CLINICAL TRIAL: NCT00640107
Title: Evaluation and Optimization of Ultrasound and/or MRI Hardware and Software in Existing SUNY Ultrasound and/or MRI Units and Newly Installed Commercially Available Units
Brief Title: Evaluation and Optimization of Ultrasound and/or MRI Hardware and Software
Status: Recruiting | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Marzieh Nezamzadeh, Diagnostic Radiology Physicist, State University of New York - Upstate Medical University
Other Study IDs: SUNYUMU 247517
Record Dates: First submitted 2008-03-12; First posted 2008-03-20 (Estimated); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: Magnetic Resonance Imaging; Ultrasound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate and optimize ultrasound and/or MRI hardware and software in both existing ultrasound/MRI units as well as in newly installed commercially available ultrasound/MRI units. The study also serves to familiarize the ultrasound/MRI technician staff with how to operate newly installed software sequences or hardware. The information obtained from this study will be utilized to optimize new software sequences and hardware that have been installed on the UMU ultrasound/MRI scanners. This will offer ultrasound/MRI technologists ample time to become familiar with the operation of new equipment. More specifically, the objectives of this study are to maximize contrast to noise (CNR) and signal to noise (SNR) ratios for new imaging sequences and hardware to obtain high quality images, maximize the potential of new machines and associated software/hardware to obtain the highest quality of images, and obtain the highest quality images in reasonable scan time to minimize patient motion.

DETAILED DESCRIPTION:
Magnetic Resonance Imaging (MRI) has been utilized for 20 years as a clinical and research tool at SUNY Upstate Medical University. Currently, there are five (5) MR (1 low-field 0.2 Tesla, 3 high-field 1.5 Tesla and 1 3.0 Tesla) units in use on the university campus. During this time, new imaging sequences and hardware including smaller more powerful magnets and faster computers have been developed that assist in the diagnosis of many disease processes. MR Angiography, MR Spectroscopy, diffusion weighted imaging and a dedicated combination Neurovascular head and neck coil are just several of the many imaging sequences and specialized coils that have been developed over the last several years.

New imaging sequences and hardware including 4.0 and 7.0 Tesla magnets are currently undergoing development and testing at several universities in the United States and worldwide. As a consequence of the many new innovations in MR imaging we must periodically upgrade our existing MR units and on occasion replace one of our existing MR units or purchase a new MR unit. This will ensure that we have the most up to date MR equipment to provide state of the art diagnostic imaging capabilities at University Hospital. The new imaging sequences and/or hardware must be optimized for each MR unit to achieve the highest signal to noise (SNR) and contrast to noise (CNR) ratios in a reasonable scan time. This practice is routinely performed at every university and private hospital as well as outpatient imaging center when a new MR unit is installed and when an existing unit is upgraded.

Ultrasound imaging has been a component of the Radiology Department since 1975 and used as a clinical and research tool. Presently our machines include the GE's models: Logic E9, S8, Logic (, P5, P6, Logic Book, Phillips IU22, SonoSite Turbo (multiple units), Siemens Acuson (x3 units) and a Siemens X300. There are updated ultrasound machines that allow color Doppler images and elastography acquisition ability. Upgrades for software and hardware are on an ongoing basis along with new applications and imaging protocols.

ELIGIBILITY:
Inclusion Criteria:

* Able to Understand and Sign Informed Consent Disclosure (ICD)
* Healthy Volunteers Aged 18-70
* Healthy Volunteers with No History of Aneurysm Clips, Cardiac Pacemakers, Claustrophobia, Neurostimulators, and Pregnancy.

Exclusion Criteria:

* Subjects > 300 Pounds
* Subjects < 18 Years Old
* Subjects > 70 Years Old
* Subjects w/ Aneurysm Clips
* Subjects w/ Cardiac Pacemakers
* Subjects w/ Claustrophobia
* Subjects w/ Neurostimulators
* Subjects w/ Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of healthy volunteers aged 18-70 who are able and willing to sign an informed consent disclosure (ICD) form to undergo an MRI scan if they meet all screening criteria.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2007-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2030-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marzieh Nezamzadeh, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data will be the only information available for sharing purposes.